CLINICAL TRIAL: NCT04791579
Title: Prophylactic Antibiotics Following Treatment of Neurogenic Overactive Bladder With Intradetrusor onabotulinumtoxinA for the Reduction of Postoperative UTI: a Randomized Blinded Placebo-controlled Trial
Brief Title: Antibiotic Prophylaxis for Neurogenic Bladder Botox
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: Pro00108452
Record Dates: First submitted 2021-03-08; First posted 2021-03-10 (Actual); Last update posted 2025-02-17 (Actual); Status verified 2025-02

CONDITIONS: Neurogenic Bladder; Post-operative Urinary Tract Infections
Keywords: prophylaxis; post-operative infection; Botox
MeSH Terms: conditions — Urinary Bladder, Neurogenic | interventions — Ciprofloxacin

STUDY DESIGN:
Intervention Model Description: Patients will be randomized at a 1:1 allocation ratio to two parallel treatment arms - intervention versus placebo
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Quadruple (Participant, Care Provider, Investigator, Outcomes Assessor) Placebo
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment Arm (Active Comparator): Ciprofloxacin 500 mg PO every 12 hrs for 3 days following the procedure
  Interventions: Drug: Ciprofloxacin
- Placebo Arm (Placebo Comparator): Placebo pill PO every 12 hrs for 3 days following the procedure
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ciprofloxacin — Fluoroquinolone antibiotic
  Arms: Treatment Arm
Drug: Placebo — Placebo pill
  Arms: Placebo Arm

SUMMARY:
Injection of Botox into the bladder is a procedure used to treat neurogenic overactive bladder at the Dianne and Irving Kipnes Urology Centre in the Kaye Edmonton Clinic. A common complication following bladder Botox is bladder infection. There are no well-studied preventative antibiotics given at the time of bladder Botox for the reduction of post-operative bladder infection. We are proposing a research study that will randomize participants into two groups - one receiving antibiotics and the other receiving placebo pills following bladder Botox. The main goal of our study is to determine if preventative antibiotics at the time of bladder Botox injection reduces post-operative bladder infection. It will provide a valuable learning opportunity for a trainee starting their academic career through working closely with established researchers across two disciplines. We hope the results of our study can ultimately be used to improve outcomes and safety for a common Urologic procedure. In addition, findings from our study could help reduce unnecessary use of antibiotics resulting in cost savings in the health care system and reduction in the risk of antibiotic resistance.

DETAILED DESCRIPTION:
This study will be a single-centred, double-blinded, randomized, placebo- controlled trial. Recruitment will be undertaken in the Urology clinic in the Urology Centre at the Kaye Edmonton Clinic in Edmonton, AB. Participants will be randomized to treatment or placebo arm with a 1:1 allocation ratio. Patients and surgeons will be blinded.

On the day of the procedure, a urine culture will be collected preoperatively to identify pre-existing bacteriuria. Technique and dose of Botox injection will be at the discretion of the operating physician. Trigone-sparing technique with injection of 200 units of Botox distributed across 10 to 20 sites is generally used at our centre.

Follow-up will occur over a six-week postoperative period. A questionnaire will be used at each follow-up encounter to screen patients for urinary tract infection symptoms, voiding dysfunction, and other adverse events potentially related to the prophylactic antibiotics. Urine cultures will be collected to confirm infection for patients developing postoperative symptoms.

ELIGIBILITY:
Inclusion Criteria:

1. Participants with neurogenic OAB, defined as OAB associated with a neurologic condition such as multiple sclerosis, Parkinson's disease, spinal cord injury, previous stroke, or any other neurologic condition the participant may have been told is a cause of their OAB symptoms
2. Age ≥ 18
3. Participants must be able to read, speak, and write in English
4. No contraindication to injection of Botox - hypersensitivity to any botulinum toxin preparation or to any of the components in the formulation, symptomatic urinary retention or PVR > 200 mL, unwillingness or inability to initiate CIC post-treatment if required.
5. No contraindication to oral Ciprofloxacin - hypersensitivity or allergy to Ciprofloxacin or other fluoroquinolone, concurrently taking Tizanidine or Agomelatine.
6. No active antibiotic therapy for any indication at the time of Botox injection
7. Not pregnant and/or breastfeeding - Botox is contraindicated in pregnancy (screen serum pregnancy test 72 hrs prior to the procedure is standard of care).
8. No active symptomatic UTI the day of the procedure - wherein the participant presents the day of their Botox procedure with new or worsening urinary frequency, urgency, dysuria, hematuria, suprapubic/flank pain, fevers or chills, will be ground for exclusion from the study - bladder Botox is contraindicated in patients with active symptomatic UTI

Exclusion Criteria:

1. Participants with idiopathic OAB
2. Age < 18
3. Patients who cannot read, speak, and write in English
4. Any contraindication to injection of Botox - hypersensitivity to any botulinum toxin preparation or to any of the components in the formulation, symptomatic urinary retention or PVR > 200 mL, unwillingness or inability to initiate CIC post-treatment if required.
5. Any contraindication to oral Ciprofloxacin - hypersensitivity or allergy to Ciprofloxacin or other fluoroquinolone, concurrently taking Tizanidine or Agomelatine.
6. Active antibiotic therapy for any indication at the time of Botox injection
7. Pregnant (as indicated by pre-operative serum quantitative B-hCG for patients aged 18 to 51 without previous hysterectomy) and/or breastfeeding
8. Active symptomatic UTI the day of the procedure - wherein the participant presents with new or worsening frequency, urgency, dysuria, hematuria, suprapubic/flank pain, fevers or chills, will be ground for exclusion from the study.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2025-02-01 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Rate of Postoperative Urinary Tract Infection | 2 weeks following the procedure
  new or worsening symptoms (dysuria, hematuria, frequency, urgency, suprapubic/flank pain, fever) AND positive urine culture (>10^5 CFU/mL)

SECONDARY OUTCOMES:
Rate of Postoperative Urinary Tract Infection | 1 and 6 weeks following the procedure
  new or worsening symptoms (dysuria, hematuria, frequency, urgency, suprapubic/flank pain, fever) AND positive urine culture (>10^5 CFU/mL)
Rate of Other Adverse Events | 1, 2 and 6 weeks following the procedure
  New onset of side effects possibly related to Ciprofloxacin (nausea/vomiting, headache, abdominal pain, constipation, diarrhea, other)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Alberta, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No